CLINICAL TRIAL: NCT02783560
Title: The Role of Sleep in Addressing Disruptive Behavior in Children
Brief Title: Behavioral Sleep Intervention in Children With Disruptive Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Indiana University School of Medicine (Other)
Responsible Party: Principal Investigator, Sarah Honaker, Assistant Professor of Pediatrics, Indiana University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2286108; UL1TR001108 (NIH)
Record Dates: First submitted 2016-05-17; First posted 2016-05-26 (Estimated); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Insomnia; Disruptive Behavior Disorder; Oppositional Defiant Disorder
Keywords: Sleep; Electrodermal Activity; Mealtimes
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Attention Deficit and Disruptive Behavior Disorders; Oppositional Defiant Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sleep First (Experimental): Families in this condition will receive a behavioral sleep intervention program (The Sleep Train Program) first, prior to a parent training intervention for disruptive behavior. After the completion of the parent training program and several assessment periods, families will receive the mealtime intervention (The Family Mealtimes Program).
  Interventions: Behavioral: The Sleep Train Program; Behavioral: The Family Mealtimes Program
- Mealtimes First (Active Comparator): Families in this active comparison condition will receive a behavioral treatment to promote positive family mealtimes first, prior to a parent training intervention for disruptive behavior. After the completion of the parent training program and several assessment periods, families will receive a behavioral sleep intervention (The Sleep Train Program).
  Interventions: Behavioral: The Sleep Train Program; Behavioral: The Family Mealtimes Program

INTERVENTIONS:
Behavioral: The Sleep Train Program — This modular behavioral sleep intervention includes required modules on sleep routines and sleep habits, and optional modules on bedtime problems, fears, anxiety, and independent sleep.
Behavioral: The Family Mealtimes Program — This modular behavioral mealtime intervention includes required modules on mealtime routines and healthy mealtime habits, and optional modules on picky eating and mealtime behavior difficulties.

SUMMARY:
Despite the high prevalence of sleep difficulties in children with disruptive behavior disorders, little is known about the role of sleep in treating disruptive behavior. The current study evaluates the addition of a sleep intervention to an existing parent-training program for caregivers of children ages 3-8 with disruptive behaviors. Objectives are to examine the impact of a novel sleep treatment program on sleep, disruptive behavior, and other measures of family functioning, utilizing a variety of self-report and objective measures (e.g. actigraphy, electrodermal activity). The investigators hypothesize that sleep intervention will result in improvements in sleep and disruptive behavior compared to control group receiving a highly plausible addition to the standard parent training intervention, and that sleep outcomes will moderate overall treatment success.

DETAILED DESCRIPTION:
Overview: The current study, which is a collaboration between Indiana University at Bloomington (PI: Bates) and Indiana University School of Medicine (PI: Honaker), seeks to evaluate the impact of adding a sleep component to a parenting intervention that has been shown to effectively treat disruptive behavior in children. A mealtime intervention will serve as an active control for the sleep treatment component, as the mealtime intervention targets changes in a family routine but is unlikely to significantly impact sleep. Participants who receive the sleep component are expected to show significant improvements in sleep compared to the mealtime group. The investigators further hypothesize that children receiving the sleep intervention will have reduced presleep arousal levels compared to baseline, and will show greater reduction in presleep arousal levels than the mealtime/control group. Finally, because of the documented links between poor sleep and externalizing behavior problems and theoretical arguments about sleep mechanisms supporting emotional and behavioral self-regulation, the investigators hypothesize that the participants who receive the sleep component will show greater reductions in disruptive behavior compared to the mealtime/control group.

Participants and Design: Participants are 3-8-year-old children who exhibit disruptive behaviors and their parents. Participants meeting criteria for the parent-training program offered as part of the general clinic practice would be approached by the therapist to discuss participation in the study. Following the consent procedure, they would be randomly assigned to one of two groups. The sleep intervention group would receive a brief, novel sleep intervention (The Sleep Train Program) in the context of the parenting program's Setting Up for Success segment, which focuses on positive routines. Sleep would be addressed briefly as needed in subsequent sessions. The mealtime/control group would not receive any particular intervention or guidance regarding sleep, but would instead focus on the routine of mealtimes. All families would then receive the same core intervention for disruptive behavior. Following the completion of the data collection, families who received the sleep component would receive the mealtime component, and vice versa.

Interventions: The existing parenting skills intervention is largely built on Troubled Families: A Treatment Program, a manualized treatment approach with extensive empirical support, selected as it is currently delivered by clinical psychology trainees at the Psychological Clinic at Indiana University in Bloomington. The sleep intervention and control intervention focusing on mealtime structure have been designed to be parallel in terms of structure and length. Though neither intervention has been evaluated (both were developed for this study), both incorporate treatment strategies with an empirical basis. The sleep intervention focuses on sufficient sleep, healthy sleep habits, and a positive bedtime routine, with optional modules to help address bedtime problems, night wakings, fears, anxiety, and independent sleep. The mealtime intervention focuses on healthy mealtime habits and mealtime routines, with optional modules to address picky eating and disruptive mealtime behaviors.

Data collection and measures: Some data will be recorded daily throughout the study, including parent diary measures of child sleep and the main child misbehaviors (noncompliance, tantrums, aggression). Other data will be collected in 4 major assessments periods. The baseline assessment will occur at the end of the initial assessment with the family and prior to the first treatment session. The midpoint assessment will occur prior to the start of the discipline intervention, approximately six week after the start of treatment. This assessment period allows for evaluation of disruptive behavior and sleep following the sleep component and an introductory segment (Setting Up for Success), but prior to the initiation of the core disruptive behavior / parenting intervention. In other words, any improvements in disruptive behavior could be attributed largely to the sleep or mealtime addition rather than the core parenting intervention. The second midpoint assessment will occur following the core intervention, but prior to initiating the sleep/mealtime component not previously covered. This allows for the evaluation of the combined sleep and disruptive behavior interventions, as well as a comparison in treatment outcomes for those who received the sleep component and those who received the mealtime/control component. A final assessment will occur following the conclusion of treatment. Survey data will be collected using on-line forms created in REDCap, and completed on a tablet that will be loaned to the family.

Measures were selected to assess sleep, disruptive behavior, child daytime functioning more generally, and family functioning. An actigraph is worn by the child for one week during each of the four assessment periods, with interpretation aided by the accompanying sleep diary. An Empatica E3 device will be used to assess electro dermal activity (EDA) as a measure of presleep arousal. The child will be asked to wear this device each evening from the start of the bedtime routine through sleep onset, at which point the parent is asked to remove the device.

Individuals collaborating on this study include: John Bates PhD (co-PI), Indiana University at Bloomington; Amy Williams PhD, Indiana University School of Medicine, and several graduate students at Indiana University in Bloomington, specifically Maureen McQuillan, Caroline Hoyniak, Brittany Rudd, and Kyle Gerst.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver participating in treatment lives at home with the child at least 50% of the time
* Child has an Eyberg Problem or Intensity T score of 60 or greater OR an Achenbach score of 60 or greater on the Externalizing scale

Exclusion Criteria:

* Child is working with another therapist or provider to address either sleep or disruptive behaviors
* Child is taking medications known to impact sleep
* Child has symptoms of obstructive sleep apnea (OSA) and OSA has not been ruled out via a sleep study
* Child has a sibling who is already participating in the study
* Child has been diagnosed with an autism spectrum disorder

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Child Externalizing Symptoms (after sleep or control/mealtime intervention) | Change from baseline (first visit) to midpoint 1 (after sleep or mealtime intervention, approximately 6 weeks after visit 1).
  Eyberg Child Behavior Inventory, Intensity Score

SECONDARY OUTCOMES:
Objective Estimate of Child Sleep Patterns (after sleep or control/mealtime intervention) | Change from baseline (first visit) to midpoint 1 (after sleep or mealtime intervention, approximately 6 weeks after visit 1).
  Actigraphy, worn by child for 1 week at each time point
Objective Estimate of Child Sleep Patterns (after sleep or control/mealtime intervention + parent training) | Change from baseline (first visit) to midpoint 2 (after parent training but before crossover, approximately 12-14 weeks after baseline)
  Actigraphy, worn by child for 1 week at each time point
Objective Estimate of Child Sleep Patterns (before and after sleep intervention; pre/post) | Change from baseline (first visit) to midpoint 1 (after sleep, approximately six weeks after visit 1) for the sleep condition and midpoint 2 to final (approximately six week after midpoint 2) for the mealtime condition.
  Actigraphy, worn by child for 1 week at each time point
Subjective Report of Child Sleep Patterns (after sleep or control/mealtime intervention) | Change from baseline (first visit) to midpoint 1 (after sleep/mealtime intervention, approximately 6 weeks after visit 1).
  Composite of two subscales ("Going to Bed" and "Falling Asleep") from the Children's Sleep Wake Scale
Subjective Report of Child Sleep Patterns (after sleep or control/mealtime intervention + parent training) | Change from baseline (first visit) to midpoint 2 (after parent training but before crossover, approximately 12-14 weeks after baseline)
  Composite of two subscales ("Going to Bed" and "Falling Asleep") from the Children's Sleep Wake Scale
Subjective Report of Child Sleep Patterns (before and after sleep intervention; pre/post) | Change from baseline (first visit) to midpoint 1 (after sleep, approximately six weeks after visit 1) for the sleep condition and midpoint 2 to final (approximately six week after midpoint 2) for the mealtime condition.
  Composite of two subscales ("Going to Bed" and "Falling Asleep") from the Children's Sleep Wake Scale
Child Externalizing Symptoms (after sleep or control/mealtime intervention + parent training) | Change from baseline (first visit) to midpoint 2 (after parent training but before crossover, approximately 12-14 weeks after baseline)
  Eyberg Child Behavior Inventory, Intensity Score
Parental Sleep (after sleep or control/mealtime intervention) | Change from baseline (first visit) to final (appoximately 3 months after visit 1).
  Actigraphy, worn by parent for 1 week at each time point
Parental Stress (before and after sleep intervention; pre/post) | Change from baseline (first visit) to midpoint 1 (after sleep, approximately 6 weeks after visit 1) for the sleep condition and midpoint 2 to final (approximately six week after midpoint 2) for the mealtime condition.
  Parenting Stress Index Short Form (PSI-4-SF)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah M Honaker, PhD, Principal Investigator — Indiana University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McQuillan ME, Bates JE, Hoyniak CP, Staples AD, Honaker SM. Children's Sleep and Externalizing Problems: A Day-to-day Multilevel Modeling Approach. Behav Sleep Med. 2023 Nov 2;21(6):712-726. doi: 10.1080/15402002.2022.2156510. Epub 2022 Dec 13. PMID 36514294